CLINICAL TRIAL: NCT01313130
Title: ADVANCED MRI IN ACUTE MILITARY TBI
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Washington University School of Medicine (Other)
Collaborators: Landstuhl Regional Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Brody, MD, PhD, Associate Professor of Neurology, Washington University School of Medicine
Other Study IDs: PT090444
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; post traumatic stress disorder; Diffusion tensor imaging; resting state functional connectivity; genetic factors
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- blast-related TBI: 100 active duty US military personnel identified clinically as having suffered blast-related TBI
- non-blast-related TBI: 100 active duty US military personnel identified clinically as having suffered non-blast-related TBI. TBI caused by other mechanisms such as motor vehicle crashes, falls, struck by blunt objects etc.
- other blast-related injuries: 100 active duty US military personnel with blast-exposure and other blast-related injuries but no clinical evidence of TBI
- other non-blast injuries: 100 active duty US military personnel with other non-blast injuries and no clinical evidence of TBI

SUMMARY:
Traumatic brain injury can cause permanent problems with thinking, memory, control of emotions, organization and planning. Thousands of soldiers, marines, and other military personnel have had injuries to the brain due the wars in Iraq and Afghanistan. Very large numbers of civilians, up to perhaps 1.5 million people per year, in the United States also have traumatic brain injuries caused by car accidents, falls, sports-related injuries or assault.

We don't know very much about traumatic brain injuries right now, but there are some important new advances in technology that may help us learn a lot more about these injuries. One such advance involves new types of MRI scans that we think will be able to show what has happened to the brain after trauma more clearly that regular scans can. The first new scan is called diffusion tensor imaging, which shows injury to the axons (the wiring of the brain). The second new scan is called resting-state functional MRI correlation analysis, which shows how well various parts of the brain are connected to each other. Importantly, the new types of scans can be done using regular scanners that we already have in every major hospital. The innovation is entirely in how the scanners are used and how the resulting pictures are analyzed on a computer after they have been taken. We have already tested these scans on some military and civilian patients with brain injury and found them to be very helpful so far. Our overall goal is to see whether these new MRI scans will be useful for active duty military personnel who have had recent traumatic brain injuries. The most important goal will be to see if the amount of injury shown on the scans be used to predict how well the patients will do overall over the next 6-12 months. A related goal will be to see whether injuries to specific parts of the brain seen by these new scans can be used to predict whether patients will be likely to have specific problems like memory loss, attention deficit, depression, or post-traumatic stress disorder. We would also like to see whether the scans could be even more useful when combined with information about genetic factors (inherited from the parents) that can be tested in the blood. Another important goal is to compare the effects of traumatic brain injuries caused by blasts or explosions with injuries from other causes, to find out what is unique about blast injury. A final goal will be to repeat the scans 6-12 months later to see whether the new MRI scans can show whether the injuries to the brain have healed, gotten worse, or stayed the same. These new scans could help with decisions about whether military personnel can return to duty, what sort of rehabilitation and treatment would benefit them most, and what family members should watch for and expect.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of blast-related TBI of any severity, as made by the LRMC TBI screening team, based on clinical history, examination, and/or clinical imaging performed as part of standard care (CT, conventional MRI). This includes participants with both primary blast and additional mechanisms of injury ("blast-plus" injury)
2. Acute injury or injuries, defined as first occurring 0-30 days prior to enrollment.
3. Ability to provide informed consent.
4. Ability to lie still in a supine position for the duration of the scan sessions, e.g. no severe claustrophobia or limiting pain from other injuries.

   Exclusion Criteria:
5. known metallic implants or metallic foreign objects.
6. known to be HIV positive
7. known to be pregnant
8. previous major traumatic brain injury
9. contraindication to MRI for medical reasons such as arrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: active duty United States military personnel
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2010-10; Primary Completion 2013-12 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Cognitive dysfunction | 6-12 months after injury
  Assessed by neuropsychological testing
Post-traumatic stress disorder | 6-12 months after injury
  Assessed using structured clinical interviews

SECONDARY OUTCOMES:
Depression | 6-12 months after injury
  Assessed using structured clinical interviews
Neurological deficits | 6-12 months after injury
  Assessed using structured neurological examinations

CONTACTS AND LOCATIONS:
Locations (2):
- Washington University, St Louis, Missouri, United States
- Landstuhl Regional Medical Center, Landstuhl, Germany

REFERENCES:
- [Result] Mac Donald CL, Johnson AM, Wierzechowski L, Kassner E, Stewart T, Nelson EC, Werner NJ, Zonies D, Oh J, Fang R, Brody DL. Prospectively assessed clinical outcomes in concussive blast vs nonblast traumatic brain injury among evacuated US military personnel. JAMA Neurol. 2014 Aug;71(8):994-1002. doi: 10.1001/jamaneurol.2014.1114. PMID 24934200